CLINICAL TRIAL: NCT01041014
Title: Cost Effectiveness of Language Services in Hospital Emergency Departments
Brief Title: Cost Effectiveness of Language Services in Hospital Emergency Departments (EDs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 55879RWJF
Record Dates: First submitted 2009-12-28; First posted 2009-12-30 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2009-12

CONDITIONS: Language Discordance
Keywords: Limited English proficiency; Cost-effectiveness; Emergency Departments; Language Discordance; Satisfaction; Limited English proficient patients; Spanish-speaking patients
MeSH Terms: conditions — Emergencies; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Professional medical interpreter (Experimental): Limited English proficient Spanish-speaking patients seen in the treatment arm were provided with the services of a professionally-trained medical interpreter to facilitate communication between the patient and emergency department staff
  Interventions: Behavioral: Professional medical interpreter
- Control, Usual Language Services (No Intervention): Patients randomized to the control arm receive the services of the emergency departments' usual language services (i.e., a telephone language line or ad hoc interpreters).

INTERVENTIONS:
Behavioral: Professional medical interpreter — All treatment interpreters were certified bilingual in Spanish and English and had completed (1) at least 40 hours of training in medical terminology, ethics, patient privacy, and basic interpreting skills; and (2) an online course in protection of human subjects.
  Arms: Professional medical interpreter

SUMMARY:
Numerous studies suggest that the use of in-person, professionally trained medical interpreters can reduce health care costs associated with diagnosing and treating patients with limited English proficiency. However, few studies have specifically addressed the question of the cost-effectiveness of language services in health care settings. This study used a randomized controlled study design to compare the cost-effectiveness of using professional interpreters with Spanish-speaking patients seen in hospital emergency departments (EDs) versus using the usual language services available to these patients. The main goal of the study was to estimate the effect that professional interpreters have on resource utilization and patient/provider satisfaction in the ED compared to the language services usually offered in these settings. Our hypothesis was that use of trained interpreters would lead to more cost-effective provision of ED services.

ELIGIBILITY:
Inclusion Criteria:

* limited English proficient (LEP) Spanish-speaking patients
* adults aged 18 or older
* LEP parents of children seen in emergency departments

Exclusion Criteria:

* cognitively impaired, comatose, or traumatized patients
* healthy volunteers
* prisoners
* hospital employees

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness of in-person interpreters versus other language services | June 2009

SECONDARY OUTCOMES:
Satisfaction with ability to communicate | June 2009

CONTACTS AND LOCATIONS:
Overall Officials: Ann D Bagchi, Ph.D., Study Director — Mathematica Policy Research; Stacy Dale, MPA, Principal Investigator — Mathematica Policy Research; Robert Eisenstein, MD, Principal Investigator — University of Medicine and Dentistry of New Jersey
Locations (2):
- United States (2):
  - CentraState Healthcare System, Freehold, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey